CLINICAL TRIAL: NCT07260617
Title: Study of the Association Between the Composition of the Gut Microbiota and Nutritional Status in Patients Treated With Chemotherapy in Digestive Oncology
Brief Title: Association Between Composition of the Gut Microbiota and Nutritional Status in Digestive Oncology
Acronym: ONCONUTRIBIOTA
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0613; 2025-A02021-48 (Other: ID-RCB)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Digestive Cancer
Keywords: oral and fecal microbiota; digestive cancer; colorectal cancer; pancreatic cancer; chemotherapy; malnutrition; microbiome
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational arm of cancer patients starting chemotherapy: During two of their routine care visits (on the day of the first chemotherapy treatment and at the end of the first cycle of chemotherapy) stool and saliva samples will be collected, completed by additional assessments including global quality of life and nutritional quality of life questionnaires, olfactory and gustatory tests, and measurements of parameters used to determine the presence of malnutrition, general health status and oncological evaluation.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — During two routine care visits - on the day of the first chemotherapy administration and at the end of the first chemotherapy cycle - stool and saliva samples will be collected. These will be complemented by additional assessments, including global and nutritional quality of life questionnaires, olfactory and gustatory tests, and measurements of parameters related to malnutrition, general health status, and oncological evaluation (including blood sampling and specific analyses based on the radiological assessments performed as part of routine care)

SUMMARY:
Nutritional status represents a crucial issue in the management of cancer patients, as between 40% and 60% of them suffer from malnutrition at the time of diagnosis. This condition worsens morbidity, increases treatment-related adverse effects, infections, and hospitalizations, and can lead to death in 10% to 20% of cases, independently of tumor progression. Anticancer treatments often exacerbate malnutrition due to their side effects, such as loss of appetite or taste alterations.

Although international guidelines (ESPEN, ESMO, ASCO) recommend a multimodal nutritional intervention combining nutritional support and physical activity. The effectiveness of these approaches varies among patients. This variability can be explained by several factors, including individual differences in dietary intake response, metabolic status, and digestive tolerance to treatments.

The intestinal and oral microbiota appear to be key cofactors in regulating these various parameters, influencing appetite, host metabolism, and intestinal absorption. Alterations in the microbiota-particularly a decrease in bacterial diversity and an increase in Candida albicans-have been associated with appetite loss and taste perception disorders, especially in patients with digestive cancers. Therefore, the intestinal microbiota constitutes a potential therapeutic and diagnostic target to improve nutritional strategies in oncology.

Interventions targeting the microbiota (such as probiotic supplementation or fecal microbiota transplantation) have already demonstrated an impact on nutritional parameters in preclinical models of malnourished cancer-bearing mice; however, clinical data remain scarce and limited.

The ONCONUTRIBIOTA-cohort study aims to characterize and investigate the oral and intestinal microbiota of patients initiating chemotherapy for digestive cancer, in relation to their nutritional status clinical characteristics and food preferences, in order to identify potential biomarkers or therapeutic targets to optimize their nutritional management.

Patients will be followed during two of their routine care visits: on the day of the first chemotherapy treatment and at the end of the first cycle of chemotherapy. During these visits, stool and saliva samples will be collected, completed by additional assessments including global quality of life and nutritional quality of life questionnaires, olfactory and gustatory tests, and measurements of parameters used to determine the presence of malnutrition, general health status and oncological evaluation.

ELIGIBILITY:
* Inclusion Criteria * :
* Adult patient
* Patient with digestive cancer, including:

  * Borderline or locally advanced pancreatic adenocarcinoma
  * Metastatic pancreatic adenocarcinoma without symptomatic peritoneal carcinomatosis
  * metastatic colon/rectal cancer without symptomatic peritoneal carcinomatosis
* Patients with an indication for chemotherapy (induction treatment or treatment of metastatic disease)
* Patients able to eat orally at the time of inclusion in the study
* Patients with a performance status (PS) score ≤2
* Patients who agree to provide stool and saliva samples
* Patients who have given their written informed consent
* Patients affiliated with the French social security system
* Exclusion Criteria :
* Pregnant or breastfeeding women
* Patients who have received antibiotics within 3 weeks prior to the first chemotherapy treatment (excluding antibiotic prophylaxis administered in the context of surgery or endoscopy).
* Individuals receiving psychiatric care that may interfere with their ability to respond to questionnaires (in the investigator's opinion)
* Persons deprived of their liberty or subject to legal protection measures (guardianship, curatorship)
* Patients participating in another interventional study with medication
* Patients who have undergone chemotherapy for another malignant tumor in the last 12 months.
* Patients with another synchronous malignant tumor, with the exception of adequately treated carcinoma in situ of the cervix or squamous cell carcinoma of the skin, or limited basal cell or squamous cell skin cancer. This cancer must then be adequately controlled.
* Patients with symptomatic brain and/or meningeal metastases.
* Patients who have undergone digestive resection (excluding appendectomy or cholecystectomy >12 months ago).
* Patients with symptomatic peritoneal carcinomatosis prior to the start of chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with chemotherapy in digestive oncology
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in fecal microbiota composition, assessed by beta-diversity (Weighted UniFrac and Bray-Curtis) based on shotgun metagenomic data, between patients with severe, moderate, or no malnutrition evaluated at V1 and V2. | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  The difference in fecal microbiota composition, measured by beta-diversity (Weighted UniFrac and Bray Curtis) from shotgun metagenomic data, between patients with severe, moderate, and no malnutrition assessed at V1 (before 1st cure of chemotherapy) and V2 (after the first cycle of chemotherapy).
  Malnutrition is defined according to GLIM recommendations by the combination of the etiological criterion of active neoplasia common to all patients included, associated with a phenotypic criterion (BMI, weight loss, sarcopenia according to a standardized method).

SECONDARY OUTCOMES:
Difference in oral microbiota composition before and after chemotherapy treatment | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  The difference in oral microbiota composition, measured by beta-diversity (Weighted UniFrac and Bray Curtis) on shotgun metagenomic data, between malnourished and non-malnourished patients (GLIM criteria) assessed at V1 (before 1st cure of chemotherapy) and V2 (after 4 cures of chemotherapy).
Variation in the taxonomic and functional composition of the oral and fecal microbiota | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Variation in the taxonomic and functional composition of the oral and fecal microbiota (analysis by beta-diversity and differential taxa and metagenomics) between V1 (before 1st cure of chemotherapy) and V2 (after 4 cures of chemotherapy).
Fecal and oral metabolomic signatures associated with malnutrition status | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Fecal and oral metabolomic signatures associated with malnutrition status Identification of fecal and oral metabolomic signatures (by LC-MS or GC-MS) associated with malnutrition status assessed at V1 (before 1st cure of chemotherapy) and V2 (after 4 cures of chemotherapy).
Correlation between taxonomic profiles and markers of nutritional status | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Correlation between taxonomic profiles (relative abundance of bacterial taxa) and markers of nutritional status (BMI, weight loss, prealbumin, albumin, CRP) at V1 and V2; calculation of Spearman's coefficient with false positive control (FDR).
Change in nutritional parameters during chemotherapy | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Change in BMI, relative weight loss, estimated nutritional intake (24-hour survey), appetite (SEFI scale), and biological markers (albumin, prealbumin, CRP) between V1 and V2.
Intra-individual variation in blood markers of nutritional status | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Intra-individual variation in markers of nutritional status (GLIM nutritional diagnosis, prealbumin, albumin) and appetite (SEFI scale) between V1 and V2, depending on the type of chemotherapy.
Change in sensory scores during chemotherapy | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Variation in sensory scores between V1 and V2, assessed using validated questionnaires (CITAS/SA-Quest, Self-reported food appreciation).
Correlation between sensory scores and nutritional status markers | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Correlation between sensory scores and nutritional status markers (GLIM criteria, albumin, SEFI) at V1 and V2 (Spearman coefficient calculation with false positive control -FDR).
Correlation between sensory scores and the composition of oral and fecal microbiota | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Correlation between sensory scores and the composition of oral and fecal microbiota at V1 and V2 (alpha/beta diversity, relative abundances of different taxa with calculation of Spearman's coefficient with false positive control -FDR).
Correlation of patients' quality of life with the composition of oral and fecal microbiota | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Correlation of patients' quality of life (EORTC QLQ-C30 questionnaire (version 3) with the composition of oral and fecal microbiota at V1 and V2 (alpha/beta diversity, relative abundances of different taxa with calculation of Spearman's coefficient with false positive control -FDR).
Correlation between sensory scores and quality of life score | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Correlation between sensory scores (CITAS/SA-Quest, Self-reported food appreciation) and quality of life score (according to EORTC QLQ-C30 (version 3)) at V1 and V2 (Spearman's coefficient calculation with false positive control -FDR).
Correlation between nutritional status markers and quality of life score | at pre-chimotherapy or after the 1st chimotherapy treatment and the end of the first cycle of chemotherapy
  Correlation between nutritional status markers (BMI, weight loss, SEFI, albumin, CRP) and quality of life score (according to EORTC QLQ-C30 (version 3)) at V1 and V2 (Spearman's coefficient calculation with false positive control -FDR).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Benech, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Edouard Herriot Hospital - medical oncology department, Lyon
  - Croix Rousse Hospital Hepatology and Gastroenterology Department, Lyon
  - Lyon Sud Hospital - Hepatology and Gastroenterology Department, Lyon